CLINICAL TRIAL: NCT02997982
Title: Feasibility and Effects on Markers in Spinal Fluid in Persons With Early Alzheimer's Disease When Treated With Valaciclovir - Open Fas II Pilot Study (VALZ-Pilot)
Brief Title: Feasibility and Effects of Valaciclovir Treatment in Persons With Early Alzheimer's Disease
Acronym: VALZ-Pilot
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hugo Lovheim (Other)
Responsible Party: Sponsor-Investigator, Hugo Lovheim, Associate professor, Umeå University
Organization: Umeå University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UmU-2016-390-31M; 2016-002317-22 (EudraCT Number)
Record Dates: First submitted 2016-12-06; First posted 2016-12-20 (Estimated); Last update posted 2020-04-03 (Actual); Status verified 2020-04

CONDITIONS: Alzheimer Disease; Mild Cognitive Impairment; Herpes Simplex
Keywords: Alzheimer's Disease; Herpes Simplex Virus; HSV; Antiviral Drugs
MeSH Terms: conditions — Alzheimer Disease; Cognitive Dysfunction; Herpes Simplex | interventions — Valacyclovir; Tablets

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Valaciclovir treatment (Experimental): Valaciclovir 500Mg Tablet
  Interventions: Drug: Valaciclovir 500Mg Tablet

INTERVENTIONS:
Drug: Valaciclovir 500Mg Tablet — Valaciclovir treatment (oral, 500 mg tablets). First week: 500 mg three times daily, second to fourth week: 1000 mg three times daily.
  Other Names: Valtrex (R)

SUMMARY:
This study investigates the effects of Valaciclovir treatment to individuals with Alzheimer's disease or Mild Cognitive Impairment of Alzheimer's Disease Type. It is an open pilot trial where 36 participants will receive 4 weeks of Valaciclovir treatment. Participants will be investigated using different measures before and after the treatment period.

DETAILED DESCRIPTION:
This study investigates the effects of valaciclovir treatment to individuals with Alzheimer's disease (AD) or Mild Cognitive Impairment of Alzheimer's Disease Type. It is an open pilot trial where 36 participants will receive 4 weeks of oral valaciclovir treatment. To find 36 persons fulfilling inclusion criteria, up to 120 persons will be screened. Important inclusion criteria are Herpes Simplex Virus (HSV) Immunoglobulin G (IgG)-positivity (HSV carriage), Apolipoprotein E allele 4 carriage and sufficient kidney function (estimated glomerular filtration rate above 30 ml/min). All participants must give their informed consent to participation.

The valaciclovir dose will be 500 mg three times daily the first week and 1000 mg three times daily week 2-4.

Participants will be investigated using different measures before and after the treatment period: Mini Mental State Examination to assess cognitive function, Cerebrospinal fluid biomarkers of Alzheimer's disease and [18F]-FHBG-PET/CT (9-[4-[18F]fluoro-3-(hydroxymethyl)butyl]guanine positron emission tomography/computed tomography)) to possibly indicate active HSV infection within the central nervous system.

ELIGIBILITY:
Inclusion Criteria:

* Man or women, age ≥ 65 years
* Ability to take a stand and to make and to sign an informed consent to participate in the study. This implies that a person with MMSE (Mini Mental State Examination) < 18 will probably not be included.
* Diagnosed with Alzheimer's disease or mild cognitive impairment due to Alzheimer's disease. At least one brain imaging examination should have been done (CT, MR, SPECT or PET/CT) and at least one objective finding should support the diagnosis beyond specific medical history. Reduced perfusion or reduced metabolism bilaterally temporally, hippocampal atrophy or pathological markers for Alzheimer's disease in cerebrospinal fluid is such findings. Persons with vascular brain disorders e.g. severe white matter changes or previous brain infarction will not be included but those with white matter changes considered normal for their age can be included.
* Positive for anti-HSV (Herpes Simplex Virus) Immunoglobulin G (IgG) in plasma, i.e. carrier of HSV.
* Hetero or Homozygote for allele 4 of gene Apolipoprotein E.
* Stable over all medication including medication for Alzheimer's disease (rivastigmine, galantamin, donepezil or memantin) for at least one month.
* No known allergy or oversensitivity against valaciclovir or aciclovir.
* Ability to independently or by support from relative or other caretaker comply to study drug.

Exclusion Criteria:

* Renal insufficiency with estimated GFR (Glomerular Filtration Rate) ≤ 30 ml/min/1.73m2
* Ongoing treatment with anticoagulants (Warfarin, low molecular heparin or other anticoagulant agents). Antiplatelet agents in recommended dose are accepted (i.e. Acetylsalicylic acid 75 mgx1)
* Life expectancy < 1 year due to other comorbidity
* Ongoing severe somatic condition that might interfere with the patients participation in the study (i.e. ongoing cancer treatment)
* Ongoing illness that makes exams in a supine position impossible (i.e. severe heart failure, severe back pain).
* Dementia diagnosis other than Alzheimer's disease, including Vascular dementia.
* Other known neurological/neurodegenerative disorder (i.e. brain tumor, MS (Multiple sclerosis), ALS (amyotrophic lateral sclerosis))
* Claustrophobia or other contraindication for doing a PET/CT scanning.
* Depression or other psychiatric illness that requires treatment (i.e. severe psychosis or other illness with equal grade of seriousness)
* Dementia or cognitive dysfunction to such extent that an informed consent is impossible to obtain, corresponding to about MMSE-SR (Mini Mental State Examination-Swedish revision) <18.
* History of substance abuse (i.e. central nervous system stimulants or alcohol). Nicotine use is accepted.
* Not willing to participate in the study.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 33 (Actual)
Dates: Start 2016-12 (Actual); Primary Completion 2020-03-04 (Actual); Study Completion 2020-03-04 (Actual)

PRIMARY OUTCOMES:
Cerebrospinal fluid (CSF) Total Tau | Baseline and treatment day 28
  Change in CSF Total Tau between samples taken before and after drug treatment

SECONDARY OUTCOMES:
Cerebrospinal fluid (CSF) Neurofilament light chain (NFL) | Baseline and treatment day 28
  Change in CSF NFL between samples taken before and after drug treatment
Cerebrospinal fluid (CSF) phosphorylated Tau (p-Tau) | Baseline and treatment day 28
  Change in CSF p-Tau between samples taken before and after drug treatment
Cerebrospinal fluid (CSF) Amyloid beta 1-42 | Baseline and treatment day 28
  Change in Amyloid beta 1-42 between samples taken before and after drug treatment
PET/CT: [18F]-FHBG accumulation within the central nervous system (CNS) | One week before drug treatment start
  Can [18F]-FHBG-PET/CT detect replicating HSV infection within the CNS?
PET/CT: Location of [18F]-FHBG accumulation | One week before drug treatment start
  Do [18F]-FHBG accumulation locate to brain areas affected in AD?
PET/CT: [18F]-FHBG accumulation | One week before and one week after drug treatment
  Change in [18F]-FHBG accumulation after, as compared to before, drug treatment
Mini Mental State Examination - Swedish Revision (MMSE-SR) | Baseline and treatment day 28
  Change in MMSE-SR scores from baseline to after drug treatment
Cerebrospinal fluid (CSF) acyclovir concentration | Treatment day 28
  Cerebrospinal fluid (CSF) acyclovir concentration
Cerebrospinal fluid (CSF) 9-carboxymethoxymethylguanine (CMMG) concentration | Treatment day 28
  Concentration of CMMG, main acyclovir metabolite
Serum acyclovir concentration | Treatment day 28
  Serum acyclovir concentration
Serum 9-carboxymethoxymethylguanine (CMMG) concentration | Treatment day 28
  Concentration of CMMG, main acyclovir metabolite
Proportion completing the [18F]-FHBG-PET/CT investigations | For the investigations one week before and one week after drug treatment
  Is [18F]-FHBG-PET/CT a feasible examination among persons with Alzheimer's disease
Proportion completing the 28 days treatment with valaciclovir at specified doses | Treatment day 28
  Feasibility of valaciclovir treatment as measured by the number of participants completing the full treatment period at the specified dose

CONTACTS AND LOCATIONS:
Overall Officials: Hugo Lövheim, M.D., Ph.D., Principal Investigator — Umeå University, Umeå, Sweden
Locations (2):
- Sweden (2):
  - Geriatric Centre, University Hospital in Umeå, Umeå, Västerbotten County
  - Memory Clinic, Uppsala University Hospital, Uppsala

IPD SHARING:
Plan to Share IPD: No